CLINICAL TRIAL: NCT03901157
Title: The Effect of Repetitive Intake of Lipids in Alginate Gel on Food Intake and Satiety
Brief Title: Repetitive Lipid Intake and Food Intake
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: NL66473.068.19
Record Dates: First submitted 2019-04-02; First posted 2019-04-03 (Actual); Last update posted 2020-02-24 (Actual); Status verified 2020-02

CONDITIONS: Satiation; Overweight and Obesity; Satiety Response
Keywords: satiety; lipids in alginate gel; food intake
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active yogurt (Experimental): Contains 120 g yogurt + 60 g oil-gel particles (containing 6 g oil) + 24 g water
  Interventions: Dietary Supplement: Yogurt A: Active
- Control yogurt (Active Comparator): Contains 120 g yogurt + 54 g empty gel particles + 6 g oil in 24 g water
  Interventions: Dietary Supplement: Yogurt B: Control

INTERVENTIONS:
Dietary Supplement: Yogurt A: Active — Free fat yogurt containing oil-filled alginate gels
  Arms: Active yogurt
Dietary Supplement: Yogurt B: Control — Free fat yogurt containing the same amount of fat as the active one, and empty alginate gels
  Arms: Control yogurt

SUMMARY:
In the present study the investigators will investigate the effect of consuming lipids inside alginate gel once a day during 4 days on food intake and satiety feelings in healthy people with overweight. All participants will receive a test yogurt that includes the oil-filled Ca-alginate gels and a control yogurt where the oil is not inside the gels.

DETAILED DESCRIPTION:
Direct infusion of lipids into different parts of the human small intestine has demonstrated to decrease food intake and subjective appetite feelings, to increase production of the satiety hormones glucagon-like peptide 1 (GLP-1), peptide YY (PYY), and cholecystokinin (CCK), and diminishes gastrointestinal (GI) motility. Amongst oils with different degree of fatty acid saturation, safflower oil (high in linoleic acid, C18:2) was found the strongest inducer of the ileal brake. When ingested orally, however, the major part of dietary lipids will be digested and absorbed in the proximal small intestine and are not likely to induce the ileal brake mechanism. Incorporating small lipid droplets into millimeter-sized calcium (Ca)-alginate gel particles has shown promising results for ileal brake activation. Oral intake of these lipid containing gels have proven to reduce food intake in humans without inducing gastrointestinal symptoms. Contrastingly, to date little is known about repetitive activation of mechanisms of satiety and the effect on food intake. It is not known whether repetitive ileal brake activation provides a stronger brake or whether this will lead to a blunted response and adaptation.

ELIGIBILITY:
Inclusion Criteria:

* Based on medical history and previous examination, no serious gastrointestinal complaints can be defined;
* Age between 18 and 65 years. This study will include healthy adult subjects (male and female);
* BMI between 25-30 kg/m2;
* Able to participate in the study, willing to give informed consent and to comply with the study procedures and restrictions;
* Weight stable over at least the last 6 months (self-admitted; ≤5% weight change).

Exclusion Criteria:

* Self-admitted milk (-protein or lactose)- allergy/intolerance;
* Self-admitted history of severe cardiovascular, respiratory, urogenital, gastrointestinal/ hepatic, haematological/immunologic, HEENT (head, ears, eyes, nose, throat), dermatological/connective tissue, musculoskeletal, metabolic/nutritional, endocrine, neurological/psychiatric diseases, allergy, major surgery and/or laboratory assessments which might limit participation in or completion of the study protocol. The severity of the disease (major interference with the execution of the experiment or potential influence on the study outcomes) will be decided and documented by the principal investigator;
* Use of medication that can influence study end-points (to be decided by medical doctor and principal investigator), including vitamin supplementation, within 14 days prior to testing;
* Administration of investigational drugs or participation in any scientific intervention study that may interfere with this study, to be decided by the principal investigator prior to the study;
* Major abdominal surgery interfering with gastrointestinal function (uncomplicated appendectomy, cholecystectomy and hysterectomy allowed, and other surgery) upon judgement of the principal investigator;
* Dieting (medically prescribed, diabetic and vegetarian);
* Pregnancy, lactation (both self-admitted);
* Excessive alcohol consumption (>20 alcoholic units per week);
* Smoking;
* Self-admitted HIV-positive state.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2019-10-21 (Actual); Primary Completion 2020-10 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Repetitive effect on ad libitum food intake | 4 days
  Food intake of ad libitum meal (kcal), as measured during lunch (based on cumulated weight reduction of the food items provided) and during a pasta dinner (also based on weight reduction of the plate assuming a homogenous meal) after 4 days of consumption of the test product.

SECONDARY OUTCOMES:
Acute effect on ad libitum food intake | 3 and 6 hours
  Food intake of ad libitum meal (kcal), as measured during lunch (based on cumulated weight reduction of the food items provided) and during a pasta dinner (also based on weight reduction of the plate assuming a homogenous meal) on the first day of consumption of the test product.
Acute vs repetitive on ad libitum food intake | 1 day and 4 days
  The food intake on the first day of consumption of the test product (acute effect) will be compared with the food intake after 4 days of consumption of the test product (repetitive effect).
Food intake in normal living setting | 2 and 3 days
  Food intake of normal living setting (kcal), as calculated from food diaries filled by participants on day 2 and day 3 of the research periods.
Feelings of satiety and GI symptoms (VAS scores) | 1 day and 4 days
  Feelings of satiety and reduce feelings of hunger, as measured on VAS scores (satiety, fullness, hunger, desire to eat, desire to snack) and occurrence and severity of gastrointestinal (GI) symptoms that orally ingested lipids in alginate gel might give, as measured on VAS scores of GI symptoms (bloating, discomfort, pain, nausea).
Energy intake compensation | 1 day and 4 days
  Percentage of energy intake compensation at lunch and dinner.

CONTACTS AND LOCATIONS:
Overall Officials: Freddy Troost, Dr., Principal Investigator — Maastricht University
Locations (1):
- Centre for Healthy Eating and Food Innovation, Venlo, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Blomain ES, Dirhan DA, Valentino MA, Kim GW, Waldman SA. Mechanisms of Weight Regain following Weight Loss. ISRN Obes. 2013 Apr 16;2013:210524. doi: 10.1155/2013/210524. eCollection 2013. PMID 24533218
- [Background] Nicklas JM, Huskey KW, Davis RB, Wee CC. Successful weight loss among obese U.S. adults. Am J Prev Med. 2012 May;42(5):481-5. doi: 10.1016/j.amepre.2012.01.005. PMID 22516488
- [Background] Sumithran P, Proietto J. The defence of body weight: a physiological basis for weight regain after weight loss. Clin Sci (Lond). 2013 Feb;124(4):231-41. doi: 10.1042/CS20120223. PMID 23126426
- [Background] van Avesaat M, Troost FJ, Ripken D, Hendriks HF, Masclee AA. Ileal brake activation: macronutrient-specific effects on eating behavior? Int J Obes (Lond). 2015 Feb;39(2):235-43. doi: 10.1038/ijo.2014.112. Epub 2014 Jun 24. PMID 24957485
- [Background] Maljaars PW, Peters HP, Kodde A, Geraedts M, Troost FJ, Haddeman E, Masclee AA. Length and site of the small intestine exposed to fat influences hunger and food intake. Br J Nutr. 2011 Nov;106(10):1609-15. doi: 10.1017/S0007114511002054. Epub 2011 Jun 7. PMID 21736790
- [Background] Alleleyn AM, van Avesaat M, Troost FJ, Masclee AA. Gastrointestinal Nutrient Infusion Site and Eating Behavior: Evidence for A Proximal to Distal Gradient within the Small Intestine? Nutrients. 2016 Feb 26;8(3):117. doi: 10.3390/nu8030117. PMID 26927170
- [Background] Spiller RC, Trotman IF, Higgins BE, Ghatei MA, Grimble GK, Lee YC, Bloom SR, Misiewicz JJ, Silk DB. The ileal brake--inhibition of jejunal motility after ileal fat perfusion in man. Gut. 1984 Apr;25(4):365-74. doi: 10.1136/gut.25.4.365. PMID 6706215
- [Background] Welch IM, Sepple CP, Read NW. Comparisons of the effects on satiety and eating behaviour of infusion of lipid into the different regions of the small intestine. Gut. 1988 Mar;29(3):306-11. doi: 10.1136/gut.29.3.306. PMID 3356362
- [Background] Ryan AT, Luscombe-Marsh ND, Saies AA, Little TJ, Standfield S, Horowitz M, Feinle-Bisset C. Effects of intraduodenal lipid and protein on gut motility and hormone release, glycemia, appetite, and energy intake in lean men. Am J Clin Nutr. 2013 Aug;98(2):300-11. doi: 10.3945/ajcn.113.061333. Epub 2013 Jun 26. PMID 23803895
- [Background] Maljaars PW, Symersky T, Kee BC, Haddeman E, Peters HP, Masclee AA. Effect of ileal fat perfusion on satiety and hormone release in healthy volunteers. Int J Obes (Lond). 2008 Nov;32(11):1633-9. doi: 10.1038/ijo.2008.166. Epub 2008 Sep 16. PMID 18794896
- [Background] Maljaars J, Romeyn EA, Haddeman E, Peters HP, Masclee AA. Effect of fat saturation on satiety, hormone release, and food intake. Am J Clin Nutr. 2009 Apr;89(4):1019-24. doi: 10.3945/ajcn.2008.27335. Epub 2009 Feb 18. PMID 19225118
- [Background] Feinle-Bisset C, Patterson M, Ghatei MA, Bloom SR, Horowitz M. Fat digestion is required for suppression of ghrelin and stimulation of peptide YY and pancreatic polypeptide secretion by intraduodenal lipid. Am J Physiol Endocrinol Metab. 2005 Dec;289(6):E948-53. doi: 10.1152/ajpendo.00220.2005. Epub 2005 Jul 5. PMID 15998659
- [Background] Maljaars PW, Peters HP, Mela DJ, Masclee AA. Ileal brake: a sensible food target for appetite control. A review. Physiol Behav. 2008 Oct 20;95(3):271-81. doi: 10.1016/j.physbeh.2008.07.018. Epub 2008 Jul 21. PMID 18692080
- [Background] Golding M, Wooster TJ, Day L, Xu M, Lundin L, Keogh J, et al. Impact of gastric structuring on the lipolysis of emulsified lipids. Soft Matter. 2011 Mar 22;7(7):3513-23.
- [Background] Smith GP. Hervey, Harris, and the parabiotic search for lipostatic signals. Appetite. 2013 Feb;61(1):97-9. doi: 10.1016/j.appet.2012.08.024. Epub 2012 Sep 13. PMID 22983368
- [Background] Corstens MN, Berton-Carabin CC, Elichiry-Ortiz PT, Hol K, Troost FJ, Masclee AAM, et al. Emulsion-alginate beads designed to control in vitro intestinal lipolysis: Towards appetite control. J Funct Foods. 2017 Jul 1;34(Supplement C):319-28.
- [Background] Dekkers BL, Kolodziejczyk E, Acquistapace S, Engmann J, Wooster TJ. Impact of gastric pH profiles on the proteolytic digestion of mixed betalg-Xanthan biopolymer gels. Food Funct. 2016 Jan;7(1):58-68. doi: 10.1039/c5fo01085c. PMID 26599197
- [Background] Sarkar A, Juan JM, Kolodziejczyk E, Acquistapace S, Donato-Capel L, Wooster TJ. Impact of Protein Gel Porosity on the Digestion of Lipid Emulsions. J Agric Food Chem. 2015 Oct 14;63(40):8829-37. doi: 10.1021/acs.jafc.5b03700. Epub 2015 Sep 29. PMID 26378382
- [Background] Li Y, Hu M, Du Y, Xiao H, McClements DJ. Control of lipase digestibility of emulsified lipids by encapsulation within calcium alginate beads. Food Hydrocoll. 2011 Jan 1;25(1):122-30
- [Background] Zhang Z, Zhang R, Zou L, Chen L, Ahmed Y, Al Bishri W, et al. Encapsulation of curcumin in polysaccharide-based hydrogel beads: Impact of bead type on lipid digestion and curcumin bioaccessibility. Food Hydrocoll. 2016 Jul 1;58:160-70.
- [Background] Rayment P, Wright P, Hoad C, Ciampi E, Haydock D, Gowland P, et al. Investigation of alginate beads for gastro-intestinal functionality, Part 1: In vitro characterisation. Food Hydrocoll. 2009 May 1;23(3):816-22.
- [Background] Wright PJ, Ciampi E, Hoad CL, Weaver AC, van Ginkel M, Marciani L, et al. Investigation of alginate gel inhomogeneity in simulated gastro-intestinal conditions using magnetic resonance imaging and transmission electron microscopy. Carbohydr Polym. 2009 Jun 10;77(2):306-15.
- [Background] Zeeb B, Saberi AH, Weiss J, McClements DJ. Retention and release of oil-in-water emulsions from filled hydrogel beads composed of calcium alginate: impact of emulsifier type and pH. Soft Matter. 2015 Mar 21;11(11):2228-36. doi: 10.1039/c4sm02791d. PMID 25646949
- [Background] Wilcox MD, Brownlee IA, Richardson JC, Dettmar PW, Pearson JP. The modulation of pancreatic lipase activity by alginates. Food Chem. 2014 Mar 1;146(100):479-84. doi: 10.1016/j.foodchem.2013.09.075. Epub 2013 Sep 20. PMID 24176371
- [Background] Corstens MN, Berton-Carabin CC, Schroën K, Viau M, Meynier A. Emulsion encapsulation in calcium-alginate beads delays lipolysis during dynamic in vitro digestion. J Funct Foods. 2018 Jul;46:394-402.
- [Background] Hoad C, Rayment P, Cox E, Wright P, Butler M, Spiller R, et al. Investigation of alginate beads for gastro-intestinal functionality, Part 2: In vivo characterisation. Food Hydrocoll. 2009 May 1;23(3):833-9.
- [Background] Hill JO, Wyatt HR, Reed GW, Peters JC. Obesity and the environment: where do we go from here? Science. 2003 Feb 7;299(5608):853-5. doi: 10.1126/science.1079857. PMID 12574618
- [Background] Rodearmel SJ, Wyatt HR, Stroebele N, Smith SM, Ogden LG, Hill JO. Small changes in dietary sugar and physical activity as an approach to preventing excessive weight gain: the America on the Move family study. Pediatrics. 2007 Oct;120(4):e869-79. doi: 10.1542/peds.2006-2927. PMID 17908743
- [Background] Almiron-Roig E, Palla L, Guest K, Ricchiuti C, Vint N, Jebb SA, Drewnowski A. Factors that determine energy compensation: a systematic review of preload studies. Nutr Rev. 2013 Jul;71(7):458-73. doi: 10.1111/nure.12048. Epub 2013 Jun 10. PMID 23815144
- [Background] Zandstra EH, Mathey MF, Graaf C, van Staveren WA. Short-term regulation of food intake in children, young adults and the elderly. Eur J Clin Nutr. 2000 Mar;54(3):239-46. doi: 10.1038/sj.ejcn.1600927. PMID 10713747
- [Background] de Graaf C, Hulshof T. Effects of weight and energy content of preloads on subsequent appetite and food intake. Appetite. 1996 Apr;26(2):139-51. doi: 10.1006/appe.1996.0012. PMID 8737166
- [Background] Blundell J, de Graaf C, Hulshof T, Jebb S, Livingstone B, Lluch A, Mela D, Salah S, Schuring E, van der Knaap H, Westerterp M. Appetite control: methodological aspects of the evaluation of foods. Obes Rev. 2010 Mar;11(3):251-70. doi: 10.1111/j.1467-789X.2010.00714.x. Epub 2010 Jan 29. PMID 20122136
- [Background] Rolls BJ, Kim S, McNelis AL, Fischman MW, Foltin RW, Moran TH. Time course of effects of preloads high in fat or carbohydrate on food intake and hunger ratings in humans. Am J Physiol. 1991 Apr;260(4 Pt 2):R756-63. doi: 10.1152/ajpregu.1991.260.4.R756. PMID 2012246
- [Background] Dar MS, Chapman WH 3rd, Pender JR, Drake AJ 3rd, O'Brien K, Tanenberg RJ, Dohm GL, Pories WJ. GLP-1 response to a mixed meal: what happens 10 years after Roux-en-Y gastric bypass (RYGB)? Obes Surg. 2012 Jul;22(7):1077-83. doi: 10.1007/s11695-012-0624-1. PMID 22419108
- [Background] Warde-Kamar J, Rogers M, Flancbaum L, Laferrere B. Calorie intake and meal patterns up to 4 years after Roux-en-Y gastric bypass surgery. Obes Surg. 2004 Sep;14(8):1070-9. doi: 10.1381/0960892041975668. PMID 15479596
- [Background] Flancbaum L, Choban PS, Bradley LR, Burge JC. Changes in measured resting energy expenditure after Roux-en-Y gastric bypass for clinically severe obesity. Surgery. 1997 Nov;122(5):943-9. doi: 10.1016/s0039-6060(97)90336-6. PMID 9369895
- [Background] Welch I, Saunders K, Read NW. Effect of ileal and intravenous infusions of fat emulsions on feeding and satiety in human volunteers. Gastroenterology. 1985 Dec;89(6):1293-7. doi: 10.1016/0016-5085(85)90645-6. PMID 4054521
- [Background] Van Citters GW, Lin HC. Ileal brake: neuropeptidergic control of intestinal transit. Curr Gastroenterol Rep. 2006 Oct;8(5):367-73. doi: 10.1007/s11894-006-0021-9. PMID 16968603
- [Background] Peters HP, Koppert RJ, Boers HM, Strom A, Melnikov SM, Haddeman E, Schuring EA, Mela DJ, Wiseman SA. Dose-dependent suppression of hunger by a specific alginate in a low-viscosity drink formulation. Obesity (Silver Spring). 2011 Jun;19(6):1171-6. doi: 10.1038/oby.2011.63. Epub 2011 Apr 21. PMID 21512509
- [Background] Solah VA, Kerr DA, Adikara CD, Meng X, Binns CW, Zhu K, Devine A, Prince RL. Differences in satiety effects of alginate- and whey protein-based foods. Appetite. 2010 Jun;54(3):485-91. doi: 10.1016/j.appet.2010.01.019. Epub 2010 Feb 6. PMID 20144671
- [Background] Odunsi ST, Vazquez-Roque MI, Camilleri M, Papathanasopoulos A, Clark MM, Wodrich L, Lempke M, McKinzie S, Ryks M, Burton D, Zinsmeister AR. Effect of alginate on satiation, appetite, gastric function, and selected gut satiety hormones in overweight and obesity. Obesity (Silver Spring). 2010 Aug;18(8):1579-84. doi: 10.1038/oby.2009.421. Epub 2009 Dec 3. PMID 19960001
- [Background] Hoad C, Rayment P, Risse V, Cox E, Ciampi E, Pregent S, et al. Encapsulation of lipid by alginate beads reduces bio-accessibility: An in vivo 13C breath test and MRI study. Food Hydrocoll. 2011 Jul 1;25(5):1190-200.
- [Background] Bourlieu C, Menard O, De La Chevasnerie A, Sams L, Rousseau F, Madec MN, Robert B, Deglaire A, Pezennec S, Bouhallab S, Carriere F, Dupont D. The structure of infant formulas impacts their lipolysis, proteolysis and disintegration during in vitro gastric digestion. Food Chem. 2015 Sep 1;182:224-35. doi: 10.1016/j.foodchem.2015.03.001. Epub 2015 Mar 6. PMID 25842331
- [Background] Zandstra EH, de Graaf C, Van Staveren WA. Influence of health and taste attitudes on consumption of low- and high-fat foods. Food Qual Prefer. 2001 Jan;12(1):75-82.
- [Background] Corstens MN, Berton-Carabin CC, de Vries R, Troost FJ, Masclee AA, Schroen K. Food-grade micro-encapsulation systems that may induce satiety via delayed lipolysis: A review. Crit Rev Food Sci Nutr. 2017 Jul 3;57(10):2218-2244. doi: 10.1080/10408398.2015.1057634. PMID 26252442
- [Background] Anderson DM, Brydon WG, Eastwood MA, Sedgwick DM. Dietary effects of sodium alginate in humans. Food Addit Contam. 1991 May-Jun;8(3):237-48. doi: 10.1080/02652039109373974. PMID 1778263
- [Background] Georg Jensen M, Kristensen M, Astrup A. Effect of alginate supplementation on weight loss in obese subjects completing a 12-wk energy-restricted diet: a randomized controlled trial. Am J Clin Nutr. 2012 Jul;96(1):5-13. doi: 10.3945/ajcn.111.025312. Epub 2012 May 30. PMID 22648709
- [Background] Corstens MN, Troost FJ, Alleleyn AME, Klaassen T, Berton-Carabin CC, Schroen K, Masclee AAM. Encapsulation of lipids as emulsion-alginate beads reduces food intake: a randomized placebo-controlled cross-over human trial in overweight adults. Nutr Res. 2019 Mar;63:86-94. doi: 10.1016/j.nutres.2018.12.004. Epub 2018 Dec 8. PMID 30824401
- [Background] EFSA Panel on Food Additives and Nutrient Sources added to Food (ANS); Younes M, Aggett P, Aguilar F, Crebelli R, Filipic M, Frutos MJ, Galtier P, Gott D, Gundert-Remy U, Kuhnle GG, Lambre C, Leblanc JC, Lillegaard IT, Moldeus P, Mortensen A, Oskarsson A, Stankovic I, Waalkens-Berendsen I, Woutersen RA, Wright M, Brimer L, Lindtner O, Mosesso P, Christodoulidou A, Horvath Z, Lodi F, Dusemund B. Re-evaluation of alginic acid and its sodium, potassium, ammonium and calcium salts (E 400-E 404) as food additives. EFSA J. 2017 Nov 10;15(11):e05049. doi: 10.2903/j.efsa.2017.5049. eCollection 2017 Nov. PMID 32625343
- [Background] Strader AD, Vahl TP, Jandacek RJ, Woods SC, D'Alessio DA, Seeley RJ. Weight loss through ileal transposition is accompanied by increased ileal hormone secretion and synthesis in rats. Am J Physiol Endocrinol Metab. 2005 Feb;288(2):E447-53. doi: 10.1152/ajpendo.00153.2004. Epub 2004 Sep 28. PMID 15454396
- [Background] Ripken D, van der Wielen N, Wortelboer HM, Meijerink J, Witkamp RF, Hendriks HF. Steviol glycoside rebaudioside A induces glucagon-like peptide-1 and peptide YY release in a porcine ex vivo intestinal model. J Agric Food Chem. 2014 Aug 20;62(33):8365-70. doi: 10.1021/jf501105w. Epub 2014 Aug 7. PMID 25062288
- [Background] van der Wielen N, van Avesaat M, de Wit NJ, Vogels JT, Troost F, Masclee A, Koopmans SJ, van der Meulen J, Boekschoten MV, Muller M, Hendriks HF, Witkamp RF, Meijerink J. Cross-species comparison of genes related to nutrient sensing mechanisms expressed along the intestine. PLoS One. 2014 Sep 12;9(9):e107531. doi: 10.1371/journal.pone.0107531. eCollection 2014. PMID 25216051
- [Background] Koopmans HS. Satiety signals from the gastrointestinal tract. Am J Clin Nutr. 1985 Nov;42(5 Suppl):1044-9. doi: 10.1093/ajcn/42.5.1044. PMID 4061357
- See also: Obesity and overweight — http://www.who.int/mediacentre/factsheets/fs311/en/